CLINICAL TRIAL: NCT04414501
Title: A Comparison of Virtual Reality Headset and Touch Screen Tablet for Minimizing Anxiety During Separation From Caregiver and Induction of Anesthesia in Children
Brief Title: Comparison of Virtual Reality to Tablet-based Distraction in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Elizabeth Ghazal, Associate Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5180036
Record Dates: First submitted 2019-08-23; First posted 2020-06-04 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-03

CONDITIONS: Anxiety, Separation
MeSH Terms: conditions — Anxiety, Separation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tablet study group (Active Comparator): Anxiety at separation from caregiver was measured by the modified Yale Preoperative Anxiety Scale (mYPAS). Caregiver anxiety was measured using the State-Trait Anxiety Inventory for Adults (STAI), a validated self-evaluation questionnaire. Mask acceptance, a functional evaluation of stress at the time of induction, was determined using the Mask Acceptance Scale.
  Interventions: Behavioral: Separation Anxiety
- VR study group (Active Comparator): Anxiety at separation from caregiver was measured by the modified Yale Preoperative Anxiety Scale (mYPAS). Caregiver anxiety was measured using the State-Trait Anxiety Inventory for Adults (STAI), a validated self-evaluation questionnaire. Mask acceptance, a functional evaluation of stress at the time of induction, was determined using the Mask Acceptance Scale.
  Interventions: Behavioral: Separation Anxiety

INTERVENTIONS:
Behavioral: Separation Anxiety — Perioperative anxiety is a common, undesirable outcome in pediatric surgical patients and has been associated with adverse outcomes.

SUMMARY:
The proposed study is a prospective randomized trial to be performed in pediatric patient's ages 4 to 10 years undergoing surgical procedures requiring general anesthesia. The purpose is to compare the effectiveness of interactive tablet devices vs. Virtual Reality headsets. The primary outcome measure being patient anxiety at the time of separation. Other comparison measures will include preoperative parent/caregiver anxiety, anesthesia mask acceptance characteristics at the time of induction, and time to fully recover in the post-operative period.

DETAILED DESCRIPTION:
After receiving IRB approval from our institution and consent from parents or guardians, ASA I or II status children ages 4 - 10 presenting for surgery requiring general anesthesia were recruited for this study. They were assigned to either tablet- or VR-based groups. At our institution, tablet-based distraction is widely used and represents standard practice. Children in this control group were given tablets in the preoperative holding area before transport to the operating room. Content consisted of entertainment apps providing access to music videos, movies and games targeting various age groups.

The study group was given a Virtual Reality Smartphone headset in the preoperative holding area prior to transport to the operating room. This headset was chosen because of its low cost and wide compatibility for a variety of smartphones. The content consisted of several VR environments that the child/parent could choose from.

In both groups, the distraction with tablet or VR was continued throughout separation from caregivers, transport to the operating room, placement of monitors and mask induction of general anesthesia. Anxiety at time of separation was measured by the modified Yale Preoperative Anxiety Scale (mYPAS). Caregiver anxiety was measured using the State-Trait Anxiety Inventory for Adults (STAI). Mask acceptance at induction of anesthesia was determined by using the Mask Acceptance Scale.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-10 years of age
* Undergoing procedure that requires general anesthesia

Exclusion Criteria:

* Emergent procedure
* ASA III-IV
* Patients with facial skin lesions
* Patients with significant history of motion sickness
* Visually impaired patients
* Patients unable to wear a virtual reality headset
* Patients receiving pharmacological intervention to decrease preoperative anxiety

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
Patient anxiety at the time of separation in children before surgical procedures | Preoperative Period
  We will compare modified Yale Preoperative Anxiety Scale (mYPAS) scores between the tablet based distraction group to those in virtual reality group. The mYPAS evaluates 27 items divided into 5 categories: activity, vocalization, emotional expressivity, state of arousal, and use of parent. The score ranges from 23 (low anxiety) to 100 (high anxiety).

SECONDARY OUTCOMES:
additional anxiety scoring techniques | Preoperative period
  Short State-Trait Anxiety Inventory for Adults (STAI). The STAI is a validated self-evaluation questionnaire measuring anxiety with scores ranging from 6 (not at all) to 24 (very much).
Mask acceptance by the patient | Intraoperative period
  Mask Acceptance Scores

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ghazal, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

REFERENCES:
- [Background] Lee J, Lee J, Lim H, Son JS, Lee JR, Kim DC, Ko S. Cartoon distraction alleviates anxiety in children during induction of anesthesia. Anesth Analg. 2012 Nov;115(5):1168-73. doi: 10.1213/ANE.0b013e31824fb469. Epub 2012 Sep 25. PMID 23011563
- [Background] Cuzzocrea F, Gugliandolo MC, Larcan R, Romeo C, Turiaco N, Dominici T. A psychological preoperative program: effects on anxiety and cooperative behaviors. Paediatr Anaesth. 2013 Feb;23(2):139-43. doi: 10.1111/pan.12100. PMID 23289773
- [Background] Esteve R, Marquina-Aponte V, Ramirez-Maestre C. Postoperative pain in children: association between anxiety sensitivity, pain catastrophizing, and female caregivers' responses to children's pain. J Pain. 2014 Feb;15(2):157-68.e1. doi: 10.1016/j.jpain.2013.10.007. Epub 2013 Oct 27. PMID 24360639
- [Background] Sheta SA, Al-Sarheed MA, Abdelhalim AA. Intranasal dexmedetomidine vs midazolam for premedication in children undergoing complete dental rehabilitation: a double-blinded randomized controlled trial. Paediatr Anaesth. 2014 Feb;24(2):181-9. doi: 10.1111/pan.12287. Epub 2013 Nov 15. PMID 24237879
- [Background] Yang KS, Habib AS, Lu M, Branch MS, Muir H, Manberg P, Sigl JC, Gan TJ. A prospective evaluation of the incidence of adverse events in nurse-administered moderate sedation guided by sedation scores or Bispectral Index. Anesth Analg. 2014 Jul;119(1):43-48. doi: 10.1213/ANE.0b013e3182a125c3. PMID 24413547
- [Background] Weiss KE, Dahlquist LM, Wohlheiter K. The effects of interactive and passive distraction on cold pressor pain in preschool-aged children. J Pediatr Psychol. 2011 Aug;36(7):816-26. doi: 10.1093/jpepsy/jsq125. Epub 2011 Jan 29. PMID 21278378
- [Background] Wohlheiter KA, Dahlquist LM. Interactive versus passive distraction for acute pain management in young children: the role of selective attention and development. J Pediatr Psychol. 2013 Mar;38(2):202-12. doi: 10.1093/jpepsy/jss108. Epub 2012 Oct 23. PMID 23092971
- [Background] Seiden SC, McMullan S, Sequera-Ramos L, De Oliveira GS Jr, Roth A, Rosenblatt A, Jesdale BM, Suresh S. Tablet-based Interactive Distraction (TBID) vs oral midazolam to minimize perioperative anxiety in pediatric patients: a noninferiority randomized trial. Paediatr Anaesth. 2014 Dec;24(12):1217-23. doi: 10.1111/pan.12475. Epub 2014 Jul 17. PMID 25040433
- [Background] Won AS, Bailey J, Bailenson J, Tataru C, Yoon IA, Golianu B. Immersive Virtual Reality for Pediatric Pain. Children (Basel). 2017 Jun 23;4(7):52. doi: 10.3390/children4070052. PMID 28644422
- [Background] Ryu JH, Park SJ, Park JW, Kim JW, Yoo HJ, Kim TW, Hong JS, Han SH. Randomized clinical trial of immersive virtual reality tour of the operating theatre in children before anaesthesia. Br J Surg. 2017 Nov;104(12):1628-1633. doi: 10.1002/bjs.10684. Epub 2017 Oct 4. PMID 28975600
- [Background] Kain ZN, Mayes LC, Cicchetti DV, Bagnall AL, Finley JD, Hofstadter MB. The Yale Preoperative Anxiety Scale: how does it compare with a "gold standard"? Anesth Analg. 1997 Oct;85(4):783-8. doi: 10.1097/00000539-199710000-00012. PMID 9322455
- [Background] Cox RG, Nemish U, Ewen A, Crowe MJ. Evidence-based clinical update: does premedication with oral midazolam lead to improved behavioural outcomes in children? Can J Anaesth. 2006 Dec;53(12):1213-9. doi: 10.1007/BF03021583. PMID 17142656
- [Background] Spielberger CD, Vagg PR. Psychometric properties of the STAI: a reply to Ramanaiah, Franzen, and Schill. J Pers Assess. 1984 Feb;48(1):95-7. doi: 10.1207/s15327752jpa4801_16. No abstract available. PMID 6707862
- [Background] Kumari S, Agrawal N, Usha G, Talwar V, Gupta P. Comparison of Oral Clonidine, Oral Dexmedetomidine, and Oral Midazolam for Premedication in Pediatric Patients Undergoing Elective Surgery. Anesth Essays Res. 2017 Jan-Mar;11(1):185-191. doi: 10.4103/0259-1162.194586. PMID 28298782
- [Background] Sikich N, Lerman J. Development and psychometric evaluation of the pediatric anesthesia emergence delirium scale. Anesthesiology. 2004 May;100(5):1138-45. doi: 10.1097/00000542-200405000-00015. PMID 15114210
- [Background] Kerimoglu B, Neuman A, Paul J, Stefanov DG, Twersky R. Anesthesia induction using video glasses as a distraction tool for the management of preoperative anxiety in children. Anesth Analg. 2013 Dec;117(6):1373-9. doi: 10.1213/ANE.0b013e3182a8c18f. PMID 24257388